CLINICAL TRIAL: NCT04023929
Title: Sources of COmplement in Meningococcal and Pertussis Serum Bactericidal Antibody Assays
Acronym: COMPAre
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.0116
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Pertussis; Meningococcal Disease; Prematurity
MeSH Terms: conditions — Whooping Cough; Meningococcal Infections; Premature Birth | interventions — Cordocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cord blood samples will be collected as part of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Term babies: Babies who are born at or after 37 gestational weeks.
  Interventions: Procedure: Cord blood sampling
- Preterm babies: Babies who are born between 32 and 36+6 gestational weeks.
  Interventions: Procedure: Cord blood sampling
- Very preterm babies: Babies who are born before 32 gestational weeks.
  Interventions: Procedure: Cord blood sampling

INTERVENTIONS:
Procedure: Cord blood sampling — A cord blood sample will be obtained after the baby has been delivered and the cord has been clamped and cut.

SUMMARY:
This study is designed to allow cord blood sample collection from the cords of babies born in three gestational age windows: ≥37 gestational weeks, 32-36+6 gestational weeks and less than 32 gestational weeks to investigate whether the result obtained using a standard hSBA assay is comparable to that achieved using complement from a gestation matched population for meningococcal B and pertussis.

DETAILED DESCRIPTION:
Newborn infants, particularly those who are born preterm, are vulnerable to infection because of their immature immune systems. Invasive meningococcal disease (IMD) and pertussis both represent significant risks to the newborn infant.

Invasive meningococcal disease (IMD), caused by Neisseria meningitidis, is a devastating illness with a case fatality rate of 10-20% even with intensive treatment. Even infants who survive IMD experience significant disability in 10-20% of cases. Serogroups A, B, C, Y, W and X cause almost all cases of IMD, and in Europe, North America and parts of Latin America serogroup B is responsible for the majority of cases. In the UK there were 747 cases of IMD in 2016/17 and Men B was responsible for 396 (53%) of these. The major burden of disease is in infants under the age of 1 year. Pertussis is a highly infectious respiratory illness caused by Bordetella pertussis which can cause significant morbidity and mortality in young infants. There has been an increase in the incidence of pertussis in the UK, along with other high income countries in recent years which has disproportionately affected young infants.

Infants in the UK are vaccinated against meningococcal group B disease at 2, 4 and 12 months with Bexsero® and against pertussis at 2,3 and 4 months as part of the 6-in-1 vaccine Infanrix hexa®. Additionally, since 2012 pregnant women in the UK have been routinely offered pertussis vaccination during pregnancy to protect the infant in the first few months of life prior to them receiving their own vaccinations.

Serum bactericidal antibody (SBA) assays are important in the assessment of immunity following vaccination and are used in the production, release and licensure of some vaccines and the evaluation of the function of others. SBA assays for pertussis and meningococcal B typically use adult complement from a healthy adult donor pool. There is some concern that using adult complement may not allow an adequate assessment of neonatal immunity. The concentration of most complement components in the neonate is around 10-80% of that in the adult and circulating regulator levels are also reduced. Differences in complement function are more pronounced in preterm infants and the differences in the quality and activation of complement in neonates raises questions about whether an SBA assay using adult complement sources allows an accurate assessment of neonatal immunity.

In this study the investigators will create a pooled complement source for three different gestational ages, ≥37 gestational weeks, 32-36+6 gestational weeks and less than 32 gestational weeks, which will allow the investigators to compare the results of the pertussis and meningococcal SBA assays when using both standard adult complement and a gestational age appropriate complement source. To do this the investigators will collect cord blood samples from deliveries within the three gestational age groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and planning to deliver at St George's University Hospitals NHS Foundation Trust

Exclusion Criteria:

* Aged less than 16 years
* Known complement deficiency

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants need to be pregnant to be recruited
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-09-21 (Estimated); Study Completion 2021-09-21 (Estimated)

PRIMARY OUTCOMES:
SBA assay results | Cord blood sampling will be performed at the time of delivery
  Comparison of the SBA assay results obtained when using adult human complement compared with a gestationally matched complement source

CONTACTS AND LOCATIONS:
Overall Officials: Anna Calvert, MBChB, Principal Investigator — St George's, Univeristy of London
Locations (1):
- St George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No